CLINICAL TRIAL: NCT00967473
Title: ACRYSOF® Toric NATURAL T9 Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-08-062
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2011-06

CONDITIONS: Bilateral Cataract
Keywords: Astigmatism; cataract; corneal astigmatism; IOL; AcrySof
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toric Intraocular Lens (Experimental): ACRYSOF® Single-Piece Toric NATURAL Intraocular Lens (IOL) Models SN60T9/SN60T8
  Interventions: Device: ACRYSOF® Single-Piece NATURAL Toric IOL Model SN60T9 and Model SN60T8.

INTERVENTIONS:
Device: ACRYSOF® Single-Piece NATURAL Toric IOL Model SN60T9 and Model SN60T8. — ACRYSOF® Single-Piece Toric NATURAL Intraocular Lens (IOL) Model SN60T9 in the first eye and either the ACRYSOF® Single-Piece Toric NATURAL IOL Model SN60T9 or Model SN60T8 in the second eye.

SUMMARY:
The purpose of this study is to describe rates of spatial distortions related to intraocular lens (IOL) misalignment for ACRYSOF® Single-Piece Toric NATURAL IOL Model SN60T9 when implanted bilaterally into the capsular bag following phacoemulsification in adult patients with bilateral cataract and regular corneal astigmatism. Subjects were implanted with the Model SN60T9 in the first operative (study) eye and either Model SN60T9 or Model SN60T8 in the second operative eye.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age or older at the time of surgery, of either gender or any race, diagnosed with bilateral cataracts;
* Calculated lens power is within the available range;
* Willing and able to complete all required postoperative visits;
* Planned cataract removal by phacoemulsification;
* Potential postoperative visual acuity of 0.2 logMAR or better in study eyes;
* Preoperative astigmatism of 4.11 - 4.62 Diopter (D) of predicted crossed cylinder as calculated by the study specific web-based Alcon® Toric IOL Calculator in the first operative eye. Corneal incisions made to reduce astigmatism will not be allowed during the course of the study;
* Preoperative astigmatism of 3.60 - 4.62 D of predicted crossed cylinder as calculated by study specific web-based Alcon® Toric IOL Calculator in the second operative eye;
* Clear intraocular media other than cataract;
* Able to comprehend and sign a statement of informed consent;
* Preoperative Best Corrected Distance Visual Acuity (BCDVA) worse than 0.2 logMAR;
* Pupil size greater than or equal to 6 mm after dilation;
* The subject must be able to undergo second eye surgery within 30 days of first eye surgery.

Exclusion Criteria:

* Irregular corneal astigmatism;
* Keratopathy/Keratectasia - any corneal abnormality, other than regular corneal astigmatism, including but not limited to the following; keratoconus, keratoglobus, keratolysis, keratomalacia, keratomycosis, and corneal plana;
* Any inflammation or edema (swelling) of the cornea, including but not limited to the following; keratitis, keratoconjunctivitis, and keratouveitis;
* Previous corneal refractive surgery;
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level worse than 0.2 logMAR;
* Amblyopia;
* Clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy);
* Diabetic retinopathy;
* Extremely shallow anterior chamber, not due to swollen cataract;
* Microphthalmos;
* Previous retinal detachment;
* Previous corneal transplant;
* Recurrent severe anterior or posterior segment inflammation of unknown etiology;
* Rubella or traumatic cataract;
* Iris neovascularization;
* Uncontrolled glaucoma;
* Aniridia;
* Optic nerve atrophy;
* Pregnancy;
* Any subject currently participating in another investigational drug or device study that may confound the results of this investigation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Toric Intraocular Lens: ACRYSOF® Single-Piece Toric NATURAL IOL Model SN60T9
Period: Overall Study
Arm/Group | Toric Intraocular Lens
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toric Intraocular Lens
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Gender [Count of Participants; unit: Participants]
  Female | 12
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Spatial Distortions Related to Intraocular Lens (IOL) Misalignment
Description: Rates of spatial distortions were evaluated by use of the Visual Distortion Questionnaire (VDQ). The VDQ evaluates the rate & frequency of subjects' experiences with potential visual distortions. The fewer the patients that report visual distortions, the better. The VDQ is a binocular assessment, therfore the subject will use both eyes to evaluate visual distortions.
Time Frame: Before Surgery and 180 days after second eye implant
Population: Per protocol, one subject was excluded from this analysis due to a secondary surgical intervention.
Measure: Number; unit: Participants
Arm/Group | Toric Intraocular Lens
Number analyzed (Participants) | 14
Participants
  Before Surgery | 11
  After Surgery | 2

2. Primary Outcome: Reduction of Cylinder
Description: Percentage of subjects with reduction in post-operative refractive cylinder (amount of astigmatism) compared to pre-operative keratometric cylinder in the study eye. The post-operative refractive cylinder should be significantly lower than it was pre-operatively.
Time Frame: 6 months after surgery on second eye
Population: All implanted subjects were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: Percent reduction of cylinder
Arm/Group | Toric Intraocular Lens
Number analyzed (Participants) | 15
Percent reduction of cylinder | 85.67 [77.04 to 94.30]

3. Primary Outcome: Lens Axis Misalignment
Description: Comparison of where the surgeon intended to place the lens axis versus final placement of the lens during the surgical procedure, measured in degrees. This number should be close to zero as there should be minimal difference between the two numbers. This assessment is only for the study eye.
Time Frame: Time of surgery
Population: All implanted subjects were included in this analysis.
Measure: Mean (Full Range); unit: Degrees
Arm/Group | Toric Intraocular Lens
Number analyzed (Participants) | 15
Degrees | 0.3 [0 to 2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Toric Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric Intraocular Lens (N=15)
Secondary Surgical Intervention (Eye disorders) | 1 (1) — One subject underwent a secondary surgical intervention (IOL repositioning) in the first eye to resolve refractive error due to inaccurate pre-operative manual keratometry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per clinical protocol confidentiality/study publication specifications all data discoveries arising out of the study, patentable of nonpatentable, shall be the sole property of Alcon Inc. Alcon reserves the right of prior review of any publication or presentation of information related to the study.